CLINICAL TRIAL: NCT00993330
Title: Macular Pigment Optical Density in Healthy Subjects
Status: Terminated | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv. - Doz. Dr, Medical University of Vienna
Other Study IDs: OPHT-310109
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Age Related Macular Degeneration
Keywords: macular pigment; to measure macular pigment in the retina
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- 1: 20 healthy subjects between 18 and 40 years
- 2: 20 healthy subjects between 41 and 50 years
- 3: 20 healthy subjects between 51 and 60 years
- 4: 20 healthy subjects between 61 and 70 years
- 5: 20 healthy subjects between 71 and 80 years
- 6: 20 healthy subjects between 81 and 90 years

SUMMARY:
The macular pigment (MP) in humans consists of the yellow, blue-absorbing carotenoids lutein and zeaxanthin, which are contained in vegetables and fruits. The highest concentrations of lutein and zeaxanthin are found in the fovea. Since light entering the eye passes through the MP before reaching the photo receptors it absorbs a significant portion of short-wavelength light. There is evidence that these absorbing properties of the MP as well as the ability of inactivating highly reactive oxygen species are protective for the retina.

Measurement of macular pigment is difficult and the investigators have recently proposed a way of measuring macular pigment optical density (MPOD) based on optical reflectometry. There is increased interest in these measurements in the recent years, because a number of studies has provided evidence that low fruit and vegetable consumption increases the risk of age related macular degeneration (AMD). The present study investigates MP optical density (OD) in healthy volunteers and is used to form a database.

Furthermore the nutritional habits and the influence on MP density will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without any signs of AMD
* Age between 18 and 90 years, (20 subjects aged between 18 and 40, 20 subjects aged between 41 and 50, 20 subjects aged between 51 and 60, 20 subjects aged between 61 and 70, 20 subjects aged between 71 and 80, 20 subjects aged between 81 and 90)
* Clear non-lenticular ocular media
* Visual acuity > 0.6

Exclusion Criteria:

* Any sign of AMD, or another retinal or optic nerve head disease
* Ocular surgery within the last 6 months
* Treatment with photosensitizing drugs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
MPOD as measured with optical reflectometry | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhofer, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria